CLINICAL TRIAL: NCT05466708
Title: Safety and Efficacy of Esketamine Combined With Dexmedetomidine for Sedation of Mechanically Ventilated Patients in the ICU: a Prospective, Randomized, Single-center Study
Brief Title: Safety and Efficacy of Esketamine Combined With Dexmedetomidine for Sedation of Mechanically Ventilated Patients
Acronym: SEEDS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021120884Esketamine
Record Dates: First submitted 2022-07-12; First posted 2022-07-20 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Dexmedetomidine; Ketamine; Analgesia; Intensive Care Units; Mechanical Ventilation
Keywords: Dexmedetomidine; Esketamine; Analgesia; Sedation; Intensive Care Units; Mechanical Ventilation
MeSH Terms: conditions — Agnosia | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esketamine combined with dexmedetomidine (Experimental): Esketamine will be administered at 1mg/kg, IVP, then intravenously pumped at 0.25-1.5mg/kg/h in combination with dexmedetomidine 1μg/kg for 20 min, followed by continuous intravenously pumped at 0.2-0.7mg/kg/h, maintaining a RASS score of -2-0.
  Interventions: Drug: Esketamine combined with dexmedetomidine
- Dexmedetomidine (Active Comparator): Dexmedetomidine will be administered at 1μg/kg for 20 min, followed by continuous intravenous pumping at 0.2-0.7mg/kg/h to maintain a RASS score of -2-0
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Esketamine combined with dexmedetomidine — Esketamine, injection, 50mg/ bottle, source: hospital pharmacy, production unit: Jiangsu Hengrui Pharmaceutical Co., LTD., validity: 2 years, storage condition: airtight shading, room temperature.
  Dexmedetomidine, injection, 0.2mg/ bottle, source: Hospital Pharmacy, manufacturer: Jiangsu Hengrui Pharmaceutical Co., LTD., expiration date: 18 months, storage condition: airtight shading, room temperature.
  Other Names: S-ketamine combined with dexmedetomidine
  Arms: Esketamine combined with dexmedetomidine
Drug: Dexmedetomidine — Dexmedetomidine, injection, 0.2mg/ bottle, source: Hospital Pharmacy, manufacturer: Jiangsu Hengrui Pharmaceutical Co., LTD., expiration date: 18 months, storage condition: airtight shading, room temperature.
  Other Names: Dexmedetomidine Hydrochloride Injection
  Arms: Dexmedetomidine

SUMMARY:
A prospective, randomized controlled study was conducted to compare the effects of esketamine combined with dexmedetomidine in the sedation and analgesia treatment of mechanically ventilated patients in the ICU on the time to awaken, time to extubation, time to mechanical ventilation, time in the ICU, and on delirium.

DETAILED DESCRIPTION:
Dexmedetomidine is a highly selective α2-adrenoceptor agonist with rapid onset of action, easy to wake up, no accumulation in the body, little inhibition of respiration, sedative, hypnotic and anxiolytic effects, and also has a certain analgesic effect.Clinical studies have shown that the use of dexmedetomidine for sedation in ICU patients is beneficial in reducing the duration of mechanical ventilation and the incidence of delirium is low, but the sedative effect of dexmedetomidine is relatively weak, and has the side effects of slowing down heart rate and lowering blood pressure, so its clinical application is limited.Esketamine is an isomer of ketamine, its effect is stronger than ketamine, and glutamate N-methyl D-aspartate (NMDA) receptor binding, play a sedative, hypnotic, analgesic effect, rapid onset, strong effect, and small respiratory inhibition, bronchodilator effect, the disadvantage is that there is a vasoconstrictor effect can cause increased blood pressure, increased heart rate.

The combination of esketamine and dexmedetomidine can provide effective sedation and analgesia with the advantages of maintaining hemodynamic stability, maintaining stable spontaneous breathing and reducing psychiatric symptoms, and has been successfully used in clinical operations such as endoscopy, pediatric anesthesia and outpatient tooth extraction.

The effectiveness and safety of esketamine in combination with dexmedetomidine for the sedation of mechanically ventilated patients in the ICU has not been evaluated. In this study, a prospective, randomized, controlled, single-center study was conducted to evaluate the efficacy and safety of esketamine in combination with dexmedetomidine for the sedation of mechanically ventilated patients in the ICU.

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated with oral endotracheal intubation in the ICU;
* Patients aged >18 years and <70 years;
* Patients with expected mechanical ventilation time >24 hours.

Exclusion Criteria:

* Known or suspected allergy to esketamine, dexmedetomidine, remifentanil, or propofol;
* Pregnancy or lactation periods;
* Obesity defined as Body Mass Index >35kg/m2;
* Extreme hemodynamic or respiratory instability due to severe burn or trauma (defined as Injury Severity Score ≥25);
* Heavy drinking defined by WHO as drinking at least 60g of pure alcohol every day for men and at least 40g for women;
* Terminally ill patients near death, such as patients with extensively metastatic tumor or refractory shock;
* Long-term exposure to sedatives, opioid analgesics or antianxiety drugs;
* Severe central nervous system disease such as cerebrovascular accidents, status epilepsy, or coma;
* Acute or chronic severe liver disease (Child-Pugh class C or history of liver transplant);
* Acute or chronic renal insufficiency needing dialysis;
* Patients or authorized surrogates refuse to provide informed consents;
* Mechanically ventilated for more than 24 hours prior to enrollment (not including the time on ventilators in the operation room).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-08-11 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Duration of mechanical ventilation | Usually within 14 days
  Duration of mechanical ventilation after endotracheal intubation

SECONDARY OUTCOMES:
Time to extubation | Usually within 14 days
  Daily offline screening, SBT test if eligible, and extubation if SBT is successful
Duration of ICU stay | Usually within 28 days
  Length of stay in ICU
28-day mortality rate | Within 28 days
  Mortality of patients within 28 days from the time of tracheal intubation
Recovery time | Within 14 days
  From the stop of sedatives to awakening
Dose of Propofol | Within 14 days
  Total dose of rescue propofol
Occurrence of delirium | Within 14 days
  The proportion of participants who have at least one positive CAM-ICU
Adverse reactions | Within 28 days
  Adverse reactions that patients experience with the medication, such as hypertension, hypotension, rapid heart rate, slow heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Zuo Xiangrong, Study Chair — Nanjing Medical University
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Zhang W, You J, Hu J, Chen X, Wang H, Li N, Wei C, Tang W, Zuo X. Effect of esketamine combined with dexmedetomidine on delirium in sedation for mechanically ventilated ICU patients: protocol for a nested substudy within a randomized controlled trial. Trials. 2024 Jul 2;25(1):431. doi: 10.1186/s13063-024-08287-3. PMID 38956664